CLINICAL TRIAL: NCT01177254
Title: Exposure to Potential Cytochrome P450 Pharmacokinetic Drug-Drug Interactions Among Osteoarthritis Patients: Incremental Risk of Multiple Prescriptions
Status: Completed | Type: Observational
Sponsor: NEMA Research, Inc. (Industry)
Responsible Party: Principal Investigator, Joseph Pergolizzi, MD, Principal Investigator, NEMA Research, Inc.
Other Study IDs: CYP450OA1
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Low Back Pain
Keywords: retrospective chronic low back pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

SUMMARY:
Using a retrospective analysis of a large commercial claims database and a Medicare database, the investigators evaluated DDEs that have the potential to cause DDIs among chronic low back pain (cLBP) patients on long-term opioid analgesia, which metabolizes through the CYP450 enzyme system, concomitant with other CYP450-metabolized drug(s).

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: retrospective chronic low back pain patients taking opioids
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)